CLINICAL TRIAL: NCT04717739
Title: Use of TTFields in Germany in Routine Clinical Care Study PROgram - Daily Activity, Sleep and Neurocognitive Functioning in Newly Diagnosed Glioblastoma Patients Study
Brief Title: TIGER PRO-Active - Daily Activity, Sleep and Neurocognitive Functioning Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 27.09.2021
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; GBM; Tumor Treating Fields; TTFields; ePRO
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- GBM with indication for TTFields: newly diagnosed GBM with clinical indication for TTFields
  Interventions: Device: TTFields

INTERVENTIONS:
Device: TTFields — Tumor Treating Fields (TTFields) help slow down or stop glioblastoma cancer cells from dividing by disrupting dividing mechanism of cancer cells leading to apoptosis. TTFields are low-intensity, intermediate frequency, alternating electric fields delivered continuously through adhesive patches, called transducer arrays, to the area of the brain where the GBM tumor is located. These transducer arrays are applied to the scalp and are connected to the wearable and portable device. TTFields are approved for the treatment of newly diagnosed and recurrent GBM.

SUMMARY:
This non-interventional study aims to investigate change over time in cognitive function, sleep quality, and activity in daily life as important determinants of QoL in a large cohort of GBM patients in Germany treated with TTFields in routine clinical care using low-threshold, electronic PRO and modern automated tracking data analyses. The gained results will allow even better understanding of TTFields therapy in daily life of GBM patients and consequently, better informing patients about what to expect when starting this therapy, increasing therapy compliance in the long-term.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common malignant primary tumor of the brain with an annual incidence of approximately 3/100.000. Since 2005 the treatment for newly diagnosed GBM consisted of maximal surgical resection, approx. 60 Gy of radiotherapy together with chemotherapy using temozolomide (TMZ), followed by 6 cycles of maintenance chemotherapy. This treatment regimen demonstrated increased median overall survival (OS) from 12.1 to 14.6 months in comparison to surgery and radiotherapy alone in 2005.

Since 2005, despite plenty of clinical phase III trials conducted, Tumor Treating Fields (TTFields) therapy was the first treatment shown to significantly increase median progression-free survival (PFS), OS and one to five year survival rates compared to the previous standard of care. These results led to FDA approval of TTFields for newly diagnosed GBM and were acknowledged since then by several guidelines recommending TTFields for GBM therapy (e.g. NCCN guidelines for CNS cancers V.1.2018, RCC guideline tumörer I hjärna och ryggmärg 2020-01-14 V3.0, DGHO guideline for glioma in adults ICD-10 C71 March 2019). Today, several national committees in Europe already list TTFields as reimbursed treatment (e.g. Austria, Sweden, Germany).

Data with TTFields therapy in real-world setting is limited and therefore further evaluation of different treatment aspects of TTFields therapy in clinical routine are of interest. In particular the QoL-related aspects neurocognitive functioning, daily activity and sleep quality in this patient cohort is of major interest, given the limited life expectancy with this disease.

This non-interventional study aims to investigate change over time in neurocognitive functioning, sleep quality, and activity in daily life as important determinants of QoL in a large cohort of GBM patients in Germany treated with TTFields in routine clinical care using low-threshold, electronic PRO and modern automated tracking data analyses. The gained results will allow even better understanding of TTFields therapy in daily life of GBM patients and consequently, better informing patients about what to expect when starting this therapy, increasing therapy compliance even further in the long-term.

ELIGIBILITY:
Inclusion Criteria:

* min.18 years of age
* Newly diagnosed, histologically confirmed GBM
* Patient after completion of radiochemotherapy but within first 3 cycles of first-line tumor-specific maintenance chemotherapy
* Clinical indication of treatment with NovoTTF-200A System (Optune®) according to IFU and medical guidelines
* Signed informed consent

Exclusion Criteria:

Any foreseeable deviation from the IFU of NovoTTF-200T Device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed, histologically confirmed GBM and an indication for treatment with NovoTTF-200A System (Optune®) according to IFU and medical guidelines will be enrolled. Patients' written informed consent to use their routine clinical data and app-based monitoring data according to data privacy standards must be obtained prior to documentation of patients' data in the e-CRF.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Time of usage of TTFields treatment in follow-up derived from monitoring data of the devices, standardised to usage days, as measure of compliance with TTFields treatment. | through study completion, an average of 18 months (mean follow-up time)
  Time of usage (compliance) of TTFields treatment over time is measured using the treatment compliance report at the Follow-up period
Number of TTFields treatment-related SAEs as assessed by the CEC standardized to one year of FU time | through study completion, an average of 18 months (mean follow-up time)
  Number of TTFields treatment-related SAEs standardized to one year of follow-up (FU) is measured using the collection of SAEs during the follow-up period
Changes in daily physical activity as a potential quality of life parameter in TTFields treatment compared to baseline for up to four months after start of TTFields therapy | Up to 4 months after start of TTFields treatment compared to baseline
  Changes in daily physical activity will be assessed by smartphone app-based clinical monitoring.
Changes in sleep quality as a potential quality of life parameter in TTFields treatment compared to baseline for up to four months after start of TTFields therapy | Up to 4 months after start of TTFields treatment compared to baseline
  Changes in sleep quality will be assessed by smartphone app-based clinical monitoring.
Changes in neurocognitive functioning as a potential quality of life parameter in TTFields treatment compared to baseline for up to four months after start of TTFields therapy. | Up to 4 months after start of TTFields treatment compared to baseline
  Changes in neurocognitive functioning will be assessed by means of MoCA interview tests.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Glas, Prof., Principal Investigator — University hospital Essen, Essen, Germany
Locations (36):
- Germany (36):
  - Universitätsklinikum Aachen, Aachen
  - Klinikum Aschaffenburg-Alzenau, Aschaffenburg
  - Universitätsklinikum Augsburg (AöR), Augsburg
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Chemnitz, Chemnitz
  - Uniklinik Köln, Cologne
  - Kliniken der Stadt Köln GmbH, Cologne
  - Carl-Thiem-Klinikum Cottbus, Cottbus
  - Universitätsklinik Carl Gustav Carus Dresden, Dresden
  - Sana Kliniken Duisburg, Duisburg
  - Universitätsklinikum Düsseldorf HHU, Düsseldorf
  - HELIOS Klinikum Erfurt, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt
  - Universitätsmedizin Greifswald, Greifswald
  - BG Klinikum Bergmannstrost Halle, Halle
  - Onkologische Schwerpunktpraxis Dres. I. Zander und E. von der Heyde, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Jena, Jena
  - Klinikum Kassel, Kassel
  - Universitätsklinikum SH Campus Kiel, Kiel
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Med. Fakultät Mannheim der Universität Heidelberg, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Klinikum Nürnberg, Nuremberg
  - Pius-Hospital Oldenburg, Oldenburg
  - Niels-Stensen-Kliniken - Marienhospital Osnabrück, Osnabrück
  - Universitätsmedizin Rostock, Rostock
  - HELIOS Kliniken Schwerin GmbH, Schwerin
  - Johanniter-Krankenhaus Genthin-Stendal GmbH, Stendal
  - Klinikum Stuttgart, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Paracelsus-Klinik Zwickau, Zwickau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostrom QT, Cioffi G, Gittleman H, Patil N, Waite K, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Other Central Nervous System Tumors Diagnosed in the United States in 2012-2016. Neuro Oncol. 2019 Nov 1;21(Suppl 5):v1-v100. doi: 10.1093/neuonc/noz150. PMID 31675094
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Stupp R, Hegi ME, Gorlia T, Erridge SC, Perry J, Hong YK, Aldape KD, Lhermitte B, Pietsch T, Grujicic D, Steinbach JP, Wick W, Tarnawski R, Nam DH, Hau P, Weyerbrock A, Taphoorn MJ, Shen CC, Rao N, Thurzo L, Herrlinger U, Gupta T, Kortmann RD, Adamska K, McBain C, Brandes AA, Tonn JC, Schnell O, Wiegel T, Kim CY, Nabors LB, Reardon DA, van den Bent MJ, Hicking C, Markivskyy A, Picard M, Weller M; European Organisation for Research and Treatment of Cancer (EORTC); Canadian Brain Tumor Consortium; CENTRIC study team. Cilengitide combined with standard treatment for patients with newly diagnosed glioblastoma with methylated MGMT promoter (CENTRIC EORTC 26071-22072 study): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2014 Sep;15(10):1100-8. doi: 10.1016/S1470-2045(14)70379-1. Epub 2014 Aug 19. PMID 25163906
- [Background] Chinot OL, Wick W, Mason W, Henriksson R, Saran F, Nishikawa R, Carpentier AF, Hoang-Xuan K, Kavan P, Cernea D, Brandes AA, Hilton M, Abrey L, Cloughesy T. Bevacizumab plus radiotherapy-temozolomide for newly diagnosed glioblastoma. N Engl J Med. 2014 Feb 20;370(8):709-22. doi: 10.1056/NEJMoa1308345. PMID 24552318
- [Background] Gilbert MR, Wang M, Aldape KD, Stupp R, Hegi ME, Jaeckle KA, Armstrong TS, Wefel JS, Won M, Blumenthal DT, Mahajan A, Schultz CJ, Erridge S, Baumert B, Hopkins KI, Tzuk-Shina T, Brown PD, Chakravarti A, Curran WJ Jr, Mehta MP. Dose-dense temozolomide for newly diagnosed glioblastoma: a randomized phase III clinical trial. J Clin Oncol. 2013 Nov 10;31(32):4085-91. doi: 10.1200/JCO.2013.49.6968. Epub 2013 Oct 7. PMID 24101040
- [Background] Stupp R, Taillibert S, Kanner AA, Kesari S, Steinberg DM, Toms SA, Taylor LP, Lieberman F, Silvani A, Fink KL, Barnett GH, Zhu JJ, Henson JW, Engelhard HH, Chen TC, Tran DD, Sroubek J, Tran ND, Hottinger AF, Landolfi J, Desai R, Caroli M, Kew Y, Honnorat J, Idbaih A, Kirson ED, Weinberg U, Palti Y, Hegi ME, Ram Z. Maintenance Therapy With Tumor-Treating Fields Plus Temozolomide vs Temozolomide Alone for Glioblastoma: A Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2535-43. doi: 10.1001/jama.2015.16669. PMID 26670971
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Gutin PH, Wong ET. Noninvasive application of alternating electric fields in glioblastoma: a fourth cancer treatment modality. Am Soc Clin Oncol Educ Book. 2012:126-31. doi: 10.14694/EdBook_AM.2012.32.122. PMID 24451721
- [Background] Gera N, Yang A, Holtzman TS, Lee SX, Wong ET, Swanson KD. Tumor treating fields perturb the localization of septins and cause aberrant mitotic exit. PLoS One. 2015 May 26;10(5):e0125269. doi: 10.1371/journal.pone.0125269. eCollection 2015. PMID 26010837
- [Background] Giladi M, Schneiderman RS, Voloshin T, Porat Y, Munster M, Blat R, Sherbo S, Bomzon Z, Urman N, Itzhaki A, Cahal S, Shteingauz A, Chaudhry A, Kirson ED, Weinberg U, Palti Y. Mitotic Spindle Disruption by Alternating Electric Fields Leads to Improper Chromosome Segregation and Mitotic Catastrophe in Cancer Cells. Sci Rep. 2015 Dec 11;5:18046. doi: 10.1038/srep18046. PMID 26658786
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Taphoorn MJB, Dirven L, Kanner AA, Lavy-Shahaf G, Weinberg U, Taillibert S, Toms SA, Honnorat J, Chen TC, Sroubek J, David C, Idbaih A, Easaw JC, Kim CY, Bruna J, Hottinger AF, Kew Y, Roth P, Desai R, Villano JL, Kirson ED, Ram Z, Stupp R. Influence of Treatment With Tumor-Treating Fields on Health-Related Quality of Life of Patients With Newly Diagnosed Glioblastoma: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2018 Apr 1;4(4):495-504. doi: 10.1001/jamaoncol.2017.5082. PMID 29392280
- [Background] Silginer M, Weller M, Stupp R, Roth P. Biological activity of tumor-treating fields in preclinical glioma models. Cell Death Dis. 2017 Apr 20;8(4):e2753. doi: 10.1038/cddis.2017.171. PMID 28425987
- [Background] Kanner AA, Wong ET, Villano JL, Ram Z; EF-11 Investigators. Post Hoc analyses of intention-to-treat population in phase III comparison of NovoTTF-100A system versus best physician's choice chemotherapy. Semin Oncol. 2014 Oct;41 Suppl 6:S25-34. doi: 10.1053/j.seminoncol.2014.09.008. Epub 2014 Sep 16. PMID 25213871
- [Background] Toms SA, Kim CY, Nicholas G, Ram Z. Increased compliance with tumor treating fields therapy is prognostic for improved survival in the treatment of glioblastoma: a subgroup analysis of the EF-14 phase III trial. J Neurooncol. 2019 Jan;141(2):467-473. doi: 10.1007/s11060-018-03057-z. Epub 2018 Dec 1. PMID 30506499
- [Background] Onken J, Goerling U, Heinrich M, Pleissner S, Krex D, Vajkoczy P, Misch M. Patient Reported Outcome (PRO) Among High-Grade Glioma Patients Receiving TTFields Treatment: A Two Center Observational Study. Front Neurol. 2019 Oct 1;10:1026. doi: 10.3389/fneur.2019.01026. eCollection 2019. PMID 31681134
- [Background] Henriksson R, Asklund T, Poulsen HS. Impact of therapy on quality of life, neurocognitive function and their correlates in glioblastoma multiforme: a review. J Neurooncol. 2011 Sep;104(3):639-46. doi: 10.1007/s11060-011-0565-x. Epub 2011 Apr 6. PMID 21468776
- [Background] Bergo E, Lombardi G, Guglieri I, Capovilla E, Pambuku A, Zagone V. Neurocognitive functions and health-related quality of life in glioblastoma patients: a concise review of the literature. Eur J Cancer Care (Engl). 2019 Jan;28(1):e12410. doi: 10.1111/ecc.12410. Epub 2015 Nov 4. PMID 26531122
- [Background] Coomans MB, Dirven L, Aaronson NK, Baumert BG, Van Den Bent M, Bottomley A, Brandes AA, Chinot O, Coens C, Gorlia T, Herrlinger U, Keime-Guibert F, Malmstrom A, Martinelli F, Stupp R, Talacchi A, Weller M, Wick W, Reijneveld JC, Taphoorn MJB. Symptom clusters in newly diagnosed glioma patients: which symptom clusters are independently associated with functioning and global health status? Neuro Oncol. 2019 Nov 4;21(11):1447-1457. doi: 10.1093/neuonc/noz118. PMID 31682733
- [Background] Armstrong TS, Shade MY, Breton G, Gilbert MR, Mahajan A, Scheurer ME, Vera E, Berger AM. Sleep-wake disturbance in patients with brain tumors. Neuro Oncol. 2017 Mar 1;19(3):323-335. doi: 10.1093/neuonc/now119. PMID 27286798